CLINICAL TRIAL: NCT02430935
Title: A Study of the Effectiveness of Cognitive Adaptation Training in Early Intervention for Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Sean Kidd, Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03/24/2015
Record Dates: First submitted 2015-04-08; First posted 2015-04-30 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Psychosis
Keywords: Psychosis; Psychosis NOS; Schizophrenia; Schizoaffective Disorder; Early Intervention
MeSH Terms: conditions — Psychotic Disorders; Mental Disorders; Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Adaptation Training (Experimental): Cognitive Adaptation Training (CAT) is a standardized approach to the use of environmental supports for improving multiple domains of adaptive functioning including adherence to medication, grooming, and activities of daily living in patients with schizophrenia.
  Interventions: Behavioral: Cognitive Adaptation Training
- Action Based Cognitive Remediation (Active Comparator): ABCR is applied in once weekly 2 hour sessions in small groups (6-8 per group). In these group sessions, simulated bridging activities are done immediately following computerized cognitive activation to increase the chance that participants retain the strategies just developed in a real life environment.
  Interventions: Behavioral: Action Based Cognitive Remediation

INTERVENTIONS:
Behavioral: Cognitive Adaptation Training — Cognitive Adaptation Training (CAT) is a manual-driven standardized approach that uses environmental supports to improve multiple domains of adaptive functioning including adherence to medication, grooming, and activities of daily living in patients with schizophrenia. Interventions for each functional deficit are based on two dimensions 1) level of impairment in executive functions (determined by neurocognitive tests) and 2) whether the overt behavior of the individual is characterized more by apathy (poverty of speech/movement/inability to initiate and follow through on behavioral sequences), disinhibition (distractibility/behavior which is highly cue-driven) or a combination of these styles (based on the Frontal Lobe Personality Scale (FLOPS).
  Arms: Cognitive Adaptation Training
Behavioral: Action Based Cognitive Remediation — ABCR is applied in once weekly 2 hour sessions in small groups (6-8 per group). In these group sessions, simulated bridging activities are done immediately following computerized cognitive activation to increase the chance that participants retain the strategies just developed in a real life environment.
  Arms: Action Based Cognitive Remediation

SUMMARY:
The proposed study will involve a randomized trial of Cognitive Adaptation Training (CAT) for early intervention as compared against an active control in which Action Based Cognitive Remediation (ABCR) will be applied.

DETAILED DESCRIPTION:
The proposed project will expand knowledge of the role of compensatory and restorative cognitive interventions for early intervention population individuals with schizophrenia. The investigators will conduct a two arm randomized trial comparing the impacts of CAT and Action Based Cognitive Remediation (ABCR) for individuals with schizophrenia who are under the age of 30. The model would mirror the investigators' preliminary work at CAMH (Kidd et al., 2014) in which there will be 4 months of specialist-delivered treatment followed by 5 months of maintenance by case managers with pre, 4 month, and 9 month evaluations conducted. This study will be among the most rigorous examinations of such interventions to date, would be among the first to examine integrative approaches, and would make a substantial contribution to the early intervention literature.

The questions for the purposes of this project are:

1. Is CAT effective among individuals with schizophrenia under the age of 30?

   and
2. Does integrating cognitive remediation with CAT enhance outcomes as compared with CAT alone?

ELIGIBILITY:
Inclusion Criteria:

* Participants must be CAMH clients, have an assigned caseworker, be between the ages of 16-34 and have a psychosis such as schizophrenia or schizoaffective disorder.

Exclusion Criteria:

* not currently experiencing high level of paranoia.

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in Adaptive Functioning (SOFAS) | Change from baseline to 4 months and 9 months
  A global level of social and occupational functioning will be obtained using the Social and Occupational Functioning Scale from the DSM-IV (American Psychiatric Association, 2000). The SOFAS rates global functioning on a scale from 0 to 100. The rating does not take into account level of symptomatology.
Change in Adaptive Functioning (SFS) | Change from baseline to 4 months and 9 months
  The Social Functioning Scale (SFS; Birchwood et al., 1990) will be administered. This is a self-report measure that details the frequency and intensity with which the person engages in functional activities. A total score and domain scores for social withdrawal, relationships, social activity, recreational activity, independence (competence), independence (performance) and employment are generated.
change in Adaptive Functioning (MCAS) | Change from baseline to 4 months and 9 months
  Both client and clinician versions of 17-item The Multnomah Community Ability Scale (MCAS, Barker et al., 1994) will be used to assess functionality.

SECONDARY OUTCOMES:
Medication Adherence | Throughout the 9 months of participation.
  Medication adherence will be determined through regular pill counts of currently prescribed psychiatric medications and pharmacy records.
Hospitalization | Throughout the 9 months of participation.
  Hospitalization will be tracked by (i) monitoring of electronic records through the central CAMH database and (ii) the reports of the primary Case Manager. Both frequency and duration of inpatient stays will be documented as will the frequency of emergency room visits.
Change in Goal Attainment (GAS) | Change from baseline to 4 months and 9 months
  Goal Attainment Scaling (GAS) will be employed as a sensitive measure of progress on individually defined goals that has demonstrated good reliability and validity with severe mental illness populations (Hurn et al., 2006). Goal attainment scaling involves the setting of 3-5 goals, each operationalized on a 5-point scale. Goals are individualized to the client and assessment of progress are determined through consensus of the clinician and case manager.
Change in Caregiver Burden (IEQ) | Change from baseline to 4 months and 9 months
  Caregiver burden will be measured for the family member involved in implementing CAT using the 31-item Involvement Evaluation Questionnaire (IEQ; Van Wijngaarden et al., 2000). This questionnaire, which has been validated for caregivers of individuals with schizophrenia, covers a broad domain of caregiving consequences and refers to burden experienced within the past 4 weeks.
Change in Cognition (WRAT-III) | Change from baseline to 4 months and 9 months
  The Wide Range Achievement Test (WRAT-III) reading subtest (Wilkinson, 1993) will be used to evaluate pre-morbid educational attainment.
Change in Cognition (Trail Making test part A) | Change from baseline to 4 months and 9 months
  The Trail Making test part A (Radford et al., 1978), a test involving using lines to connect numbers, will be used to assess scanning ability and psychomotor speed.
Change in Cognition (Digit Span Subtest of the Weschler Adult Intelligence Scale - III ) | Change from baseline to 4 months and 9 months
  Short term memory will be evaluated with the digit span subtest of the Weschler Adult Intelligence Scale - III (The Psychological Corporation, 1997).
Change in Cognition (CVLT) | Change from baseline to 4 months and 9 months
  Verbal learning and memory will be assessed with the California Verbal Learning Test (CVLT -Delis et al., 1987). The CVLT involves the repeated presentation of a word list that determines acquisition ability and retention.
Change in Cognition (Trail Making Test, Part B, and the Wisconsin Card Sorting Test) | Change from baseline to 4 months and 9 months
  Executive functioning will be assessed with the Trail Making Test, Part B, and the Wisconsin Card Sorting Test (WCST - Berg, 1948).
Change in Positive symptoms (BPRS-E) | Change from baseline to 4 months and 9 months
  Positive symptoms will be assessed using the expanded version of the Brief Psychiatric Rating Scale (BPRS-E; Ventura et al., 1993). The BPRS-E is a 24-item scale assessing multiple domains of psychopathology on a series of 7-point scales (1-7). A positive symptom factor score is composed of items assessing hallucinations, unusual thought content, conceptual disorganization and suspiciousness.
Change in Negative symptoms (NSA) | Change from baseline to 4 months and 9 months
  Negative symptoms will be assessed using the Negative Symptom Assessment (NSA; Alphs et al., 1989). The NSA is a 26-item instrument examining negative symptomatology on a series of 7-point scales (0-6). A total negative symptom score is calculated by adding together the scores from the NSA subscales, communication, emotion, motivation, social functioning, and cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Kidd, Principal Investigator — Clinician Scientist
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Alphs LD, Summerfelt A, Lann H, Muller RJ. The negative symptom assessment: a new instrument to assess negative symptoms of schizophrenia. Psychopharmacol Bull. 1989;25(2):159-63. No abstract available. PMID 2602512
- [Background] BERG EA. A simple objective technique for measuring flexibility in thinking. J Gen Psychol. 1948 Jul;39:15-22. doi: 10.1080/00221309.1948.9918159. No abstract available. PMID 18889466
- [Background] Birchwood M, Smith J, Cochrane R, Wetton S, Copestake S. The Social Functioning Scale. The development and validation of a new scale of social adjustment for use in family intervention programmes with schizophrenic patients. Br J Psychiatry. 1990 Dec;157:853-9. doi: 10.1192/bjp.157.6.853. PMID 2289094
- [Background] Delis, D., Kramer, J., Kaplan. E., & Ober, B. (1987). California Verbal Learning and Memory Test (Manual). San Antonio, TX: Psychological Corporation.
- [Background] Draper ML, Stutes DS, Maples NJ, Velligan DI. Cognitive adaptation training for outpatients with schizophrenia. J Clin Psychol. 2009 Aug;65(8):842-53. doi: 10.1002/jclp.20612. PMID 19521972
- [Background] Kelland DZ, Lewis RF. The Digit Vigilance Test: reliability, validity, and sensitivity to diazepam. Arch Clin Neuropsychol. 1996;11(4):339-44. PMID 14588938
- [Background] Kidd SA, Kaur J, Virdee G, George TP, McKenzie K, Herman Y. Cognitive remediation for individuals with psychosis in a supported education setting: a randomized controlled trial. Schizophr Res. 2014 Aug;157(1-3):90-8. doi: 10.1016/j.schres.2014.05.007. Epub 2014 Jun 2. PMID 24893903
- [Background] Kidd SA, Herman Y, Barbic S, Ganguli R, George TP, Hassan S, McKenzie K, Maples N, Velligan D. Testing a modification of cognitive adaptation training: streamlining the model for broader implementation. Schizophr Res. 2014 Jun;156(1):46-50. doi: 10.1016/j.schres.2014.03.026. Epub 2014 Apr 29. PMID 24794880
- [Background] Radford LM, Chaney EF, O'Leary MR, O'Leary DE. Screening for cognitive impairment among inpatients. J Clin Psychiatry. 1978 Sep;39(9):712-5. PMID 690089
- [Background] The Psychological Corporation. (1997). WAIS-III administration and scoring manual. San Antonio, TX: Psychological Corporation.
- [Background] Ventura J, Green MF, Shaner A, Liberman RP: Training and quality assurance with the brief psychiatric rating scale: The drift busters. International Journal of Methods in Psychiatric Research 1993; 3:221-24
- [Background] Wilkinson ,G. (1993). Wide Range Achievement Test 3 (Manual). Wilmington, DE: Wide Range Inc.
- [Background] Diagnostic and statistical manual of mental disorders (4th ed.). American Psychiatric Association, Washington, DC
- [Background] Barker S, Barron N, McFarland BH, Bigelow DA. A community ability scale for chronically mentally ill consumers: Part I. Reliability and validity. Community Ment Health J. 1994 Aug;30(4):363-83. doi: 10.1007/BF02207489. PMID 7956112
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addictions teaching hospital. — http://www.camh.ca/en/research/Pages/research.aspx